CLINICAL TRIAL: NCT02183584
Title: An Open Label, Two-period, Fixed Sequence, Phase 1 Trial to Evaluate the Effect of Multiple Doses of Rifampicin on the Multiple-dose Pharmacokinetics of Linagliptin
Brief Title: Study to Evaluate the Effect of Multiple Doses of Rifampicin on the Multiple-dose Pharmacokinetics of Linagliptin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1218.67
Record Dates: First submitted 2014-07-07; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Rifampin; Linagliptin

ARMS (1):
- Rifampicin and Linagliptin (Experimental)
  Interventions: Drug: Rifampicin; Drug: Linagliptin

INTERVENTIONS:
Drug: Rifampicin
Drug: Linagliptin

SUMMARY:
Investigation of the bioavailability of linagliptin after concomitant multiple oral administration of 5 mg linagliptin tablets and 600 mg rifampicin (Treatment A) in comparison to multiple oral administration of 5 mg linagliptin tablets given alone (Treatment B)

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), clinical laboratory tests
* Age 18 to 50 years (incl.)
* BMI 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good clinical practice (GCP) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic (incl. porphyrias), renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts.
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (more than 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (more than 10 cigarettes or more than 3 cigars or more than 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 30 g/day if male, more than 20 g/day if female)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* Thrombocytopenia or increased liver function tests (i.e. Alanine transaminase (ALT), Aspartate transaminase (AST), bilirubin, Alkaline phosphatase (AP), Gamma-glutamyl transferase (GGT)) at screening
* prior rifampicin exposure

For female subjects:

* Positive pregnancy test, pregnancy or planning to become pregnant during the study or within 2 months after study completion
* No adequate contraception during the study and until 1 month after study completion, i.e. not any of the following: IUD (intrauterine device), sexual abstinence for at least 1 month prior to enrolment, vasectomised partner (vasectomy performed at least 1 year prior to enrolment), or surgical sterilisation (including hysterectomy). Females, who do not have a vasectomised partner, are not sexually abstinent or surgically sterile have to use an additional barrier method (e.g. condom, diaphragm with spermicide)
* Lactation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-09; Primary Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Area under the steady state concentration-time curve of linagliptin in plasma (AUCτ,ss) | up to 19 days
Maximum measured steady state concentration of linagliptin in plasma (Cmax,ss) | up to 19 days

SECONDARY OUTCOMES:
Dipeptidyl-peptidase 4 (DPP-4) inhibition | up to 19 days
AUCτ,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) of CD 1790 | up to 19 days
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) of CD 1790 | up to 19 days
Ratio of urinary concentrations of 6β-hydroxycortisol to cortisol | screening, days 1 and 6 of treatment A, days 4, 6, 8 and 12 of treatment B always in the morning before drug administration
Aet1-t2,ss ( amount of analyte that is eliminated in urine from the time point t1 to time point t2 under steady state conditions) of linagliptin | up to 19 days
fet1-t2,ss ( fraction of administered drug excreted unchanged in urine at steady state over the respective time interval, where t1 and t2 define beginning and end times of the time interval) of linagliptin | up to 19 days
Number of patients with adverse events | up to 42 days
Assessment of global tolerability by investigator on a 4-point scale | up to 21 days after last drug administration
Number of patients with abnormal findings in physical examination | up to 21 days after last drug administration
Number of patients with abnormal changes in laboratory parameters | up to 21 days after last drug administration
Number of patients with clinically significant changes in Vital signs (Blood Pressure (BP), Pulse Rate (PR)) | up to 21 days after last drug administration
Number of patients with clinically significant changes in 12-lead ECG (electrocardiogram) | up to 21 days after last drug administration